CLINICAL TRIAL: NCT06289075
Title: Prognostication of ICU- and Ventilator- Days Over the Next Years Until 2040 Using Statistical Projection Models and Retrospective Data From International Databases From 2005-2023 (PrognostICate- Study).
Brief Title: PrognostICate- Study:Prognostication of ICU- and Ventilator- Days Over the Next Years Until 2040
Acronym: PrognostICate
Status: Recruiting | Type: Observational
Sponsor: University Hospital of Cologne (Other)
Collaborators: Johann Wolfgang Goethe University Hospital (Other); Monash University (Other); The Alfred (Other); Albert Einstein College of Medicine (Other)
Responsible Party: Principal Investigator, Sandra Emily Stoll, MD, Attending Anesthesiology and Intensive Care Medicine, University Hospital of Cologne
Other Study IDs: 23-1096-retro
Record Dates: First submitted 2024-02-24; First posted 2024-03-01 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: ICU Admission
Keywords: Length of ICU stay; Length of mechanical ventilation
MeSH Terms: interventions — Intensive Care Units; Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ICU patients: All ICU patients in different countries worldwide from 2005-2023
  Interventions: Other: Intensive Care Unit (ICU) treatment

INTERVENTIONS:
Other: Intensive Care Unit (ICU) treatment — ICU treatment
  Other Names: ICU treatment

SUMMARY:
The Objective of this retrospective multicenter- study is to forecast Intensive Care Unit (ICU) length of stay (ICULOS) and length of mechanical ventilation (LOMV) in ICU patients of different groups (regarding gender, age group, medical vs surgical admission) worldwide for the next years up to the year of 2040 using statistical forecasting models and historical, national and international ICU databases and population databases.

DETAILED DESCRIPTION:
Adequate resource allocation in Intensive Care Medicine is especially challenging due to limited resources and increasing demands for ICU capacities due to an aging population and medical advances. Several studies in the past were trying to predict ICULOS using different models. The Objective and aim of our retrospective multicenter study are to forecast ICU length of stay (ICULOS) and length of mechanical ventilation (LOMV) in ICU patients of different groups (regarding gender, age group, medical vs surgical admission) worldwide for the next years up to the year of 2040 using statistical forecasting models.

To achieve this objective, historical ICU data spanning from 2005 to 2023 is collected from international ICU databases worldwide as well as population data from national and international databases and employ different statistical forecasting models (ARIMA-Model (Auto-Regressive Integrated Moving Average), logistic regression, Poisson Regression and ETS (Exponential smoothing)) to make these predictions. The Validity of the 4 different models is assessed with out-of-time-cross validity by splitting the data in 2 subsets for generation and testing of the model in a ratio of approximately 75:25 of the dataset. The most valid model of the 4 different models will be chosen. The statistical analysis follows he guidelines for Accurate and Transparent Health Estimates Reporting (GATHER Statement) von Stevens et al. from the year 2016.

The ultimate goal of this project is to provide valuable insights to healthcare system decision-makers worldwide regarding future requirements of ICU beds and ventilator capacities. With this insight we want to enable healthcare- system decision makers worldwide to proactively anticipate and allocate appropriate ICU resources for the future.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to an ICU between the years 2005-2023

Exclusion Criteria:

* Patients without ICU admission or ICU admission < 4 hours

Ages: 1 Day to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: ICU patients worldwide
Sampling Method: Probability Sample
Enrollment: 10000000 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Length of mechanical ventilation | 2024-2040
  Forecasting mechanical ventilation for the next 16 years
Length of ICU stay | 2024-2040
  Forecasting ICU stay for the next 16 years

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Intensive Care Medicine, Cologne, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No